CLINICAL TRIAL: NCT00572507
Title: A Historically-controlled Single-arm Multi-center Prospective Trial to Evaluate the Safety and Efficacy of Aesculap MonoMax® Suture Material for Abdominal Wall Closure After Primary Median Laparotomy
Brief Title: Multi-center Study to Evaluate the Safety and Efficacy of Aesculap MonoMax® for Abdominal Wall Closure
Acronym: ISSAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAG-G-H-0701
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Primary Median Laparotomy
Keywords: Absorbable Monofilament Suture Material; Safety and Efficacy; Abdominal Wall/ Fascia; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MonoMax (Experimental): MonoMax is used for abdominal wall closure
  Interventions: Device: MonoMax®

INTERVENTIONS:
Device: MonoMax® — Abdominal wall closure with ultra-longterm absorbable monofilament suture after primary median laparotomy
  Other Names: ultra-longterm-absorbable monofilament suture Aesculap MonoMax®

SUMMARY:
MonoMax will be used for a continuous all-layer (except skin) suture to close abdominal wall after midline incision. The primary objective of this trial is to demonstrate that the frequency of wound infection and the frequency of reoperation due to burst-abdomen after primary median laparotomy for elective surgical intervention are equal or lower than in the INSECT trial. The secondary objectives are to demonstrate that the length of postoperative hospital stay and the frequency of abdominal hernias 12 months after the surgery are equal or lower than in the INSECT trial. [Knaebel HP et al., 2005]

ELIGIBILITY:
Inclusion Criteria:

* Age equal or greater than 18 years
* Expected survival time > 12 months
* Patient undergoing elective and primary median laparotomy
* BMI < 35
* Expected length of skin incision > 15 cm

Exclusion Criteria:

* Peritonitis
* Emergency surgery
* Coagulopathy
* Current immunosuppressive therapy (> 40 mg of a Corticoid per day or Azathioprin)
* Chemotherapy within 2 weeks before operation
* Radiotherapy of the abdomen completed less than 8 weeks before operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
frequency of wound infection, frequency of reoperation due to burst-abdomen after primary median laparotomy | till day of discharge

SECONDARY OUTCOMES:
length of postoperative hospital stay after surgery and frequency of incisional hernias 12 months after the surgery and frequency of wound infections 30 days postoperative | different

CONTACTS AND LOCATIONS:
Overall Officials: Markus W Buechler, Prof. Dr., Principal Investigator — Universitaetsklinikum Heidelberg; Chirugische Klinik; Karl-Walter Jauch, Prof. Dr., Principal Investigator — Klinikum der Universitaet Muenchen, Grosshadern; Chirurgische Klinik und Poliklinik; Annette Franck, Dr., Principal Investigator — Universitaets-Klinikum Giessen-Marburg; Klinik fuer Viszeral-, Thorax- und Gefaesschirurgie; Christoph Seidlmayer, Dr., Principal Investigator — St. Bonifatius Hospital, Lingen
Locations (4):
- Germany (4):
  - Universitaetsklinikum Heidelberg, Heidelberg
  - St. Bonifatius-Hospital; Chirurgische Klinik, Lingen
  - Universitaetsklinikum Giessen-Marburg, Klinik fuer Viszeral-, Thorax- und Gefaesschirurgie, Marburg
  - Universitaetsklinikum Muenchen Grosshadern, München

REFERENCES:
- [Background] Amgwerd M, Decurtins M, Largiader F. [Hernia of the surgical scar--predisposition or inadequate suture technique?]. Helv Chir Acta. 1992 Aug;59(2):345-8. No abstract available. German. PMID 1428925
- [Background] Eisner L, Harder F. [Incisional hernias]. Chirurg. 1997 Apr;68(4):304-9. doi: 10.1007/s001040050193. German. PMID 9206624
- [Background] Zimmermann G, Muller G, Haid A. [Surgical therapy of incisional hernias]. Chirurg. 1991 Sep;62(9):656-62. No abstract available. German. PMID 1748022
- [Background] Luijendijk RW, Lemmen MH, Hop WC, Wereldsma JC. Incisional hernia recurrence following "vest-over-pants" or vertical Mayo repair of primary hernias of the midline. World J Surg. 1997 Jan;21(1):62-5; discussion 66. doi: 10.1007/s002689900194. PMID 8943179
- [Background] Manninen MJ, Lavonius M, Perhoniemi VJ. Results of incisional hernia repair. A retrospective study of 172 unselected hernioplasties. Eur J Surg. 1991 Jan;157(1):29-31. PMID 1675878
- [Background] Paul A, Lefering R, Kohler L, Eypasch E. [Current practice of incisional hernia reconstruction in Germany]. Zentralbl Chir. 1997;122(10):859-61. German. PMID 9446447
- [Background] Paul A, Korenkov M, Peters S, Fischer S, Holthausen U, Kohler L, Eypasch E. [Mayo duplication in treatment of incisional hernia of the abdominal wall after conventional laparotomy. Results of a retrospective analysis and comparison with the literature]. Zentralbl Chir. 1997;122(10):862-70. German. PMID 9446448
- [Background] Cassar K, Munro A. Surgical treatment of incisional hernia. Br J Surg. 2002 May;89(5):534-45. doi: 10.1046/j.1365-2168.2002.02083.x. PMID 11972542
- [Background] Klinge U, Conze J, Limberg W, Brucker C, Ottinger AP, Schumpelick V. [Pathophysiology of the abdominal wall]. Chirurg. 1996 Mar;67(3):229-33. German. PMID 8681695
- [Background] Irvin TT, Stoddard CJ, Greaney MG, Duthie HL. Abdominal wound healing: a prospective clinical study. Br Med J. 1977 Aug 6;2(6083):351-2. doi: 10.1136/bmj.2.6083.351. PMID 329940
- [Background] Osther PJ, Gjode P, Mortensen BB, Mortensen PB, Bartholin J, Gottrup F. Randomized comparison of polyglycolic acid and polyglyconate sutures for abdominal fascial closure after laparotomy in patients with suspected impaired wound healing. Br J Surg. 1995 Aug;82(8):1080-2. doi: 10.1002/bjs.1800820824. PMID 7648158
- [Background] Gys T, Hubens A. A prospective comparative clinical study between monofilament absorbable and non-absorbable sutures for abdominal wall closure. Acta Chir Belg. 1989 Sep-Oct;89(5):265-70. PMID 2530745
- [Background] Bucknall TE, Ellis H. Abdominal wound closure--a comparison of monofilament nylon and polyglycolic acid. Surgery. 1981 Jun;89(6):672-7. PMID 6264641
- [Background] Israelsson LA, Jonsson T, Knutsson A. Suture technique and wound healing in midline laparotomy incisions. Eur J Surg. 1996 Aug;162(8):605-9. PMID 8891617
- [Background] Leaper DJ, Allan A, May RE, Corfield AP, Kennedy RH. Abdominal wound closure: a controlled trial of polyamide (nylon) and polydioxanone suture (PDS). Ann R Coll Surg Engl. 1985 Sep;67(5):273-5. PMID 3931536
- [Background] Wissing J, van Vroonhoven TJ, Schattenkerk ME, Veen HF, Ponsen RJ, Jeekel J. Fascia closure after midline laparotomy: results of a randomized trial. Br J Surg. 1987 Aug;74(8):738-41. doi: 10.1002/bjs.1800740831. PMID 3307992
- [Background] Cameron AE, Parker CJ, Field ES, Gray RC, Wyatt AP. A randomised comparison of polydioxanone (PDS) and polypropylene (Prolene) for abdominal wound closure. Ann R Coll Surg Engl. 1987 May;69(3):113-5. PMID 3111339
- [Background] van 't Riet M, Steyerberg EW, Nellensteyn J, Bonjer HJ, Jeekel J. Meta-analysis of techniques for closure of midline abdominal incisions. Br J Surg. 2002 Nov;89(11):1350-6. doi: 10.1046/j.1365-2168.2002.02258.x. PMID 12390373
- [Background] Hsiao WC, Young KC, Wang ST, Lin PW. Incisional hernia after laparotomy: prospective randomized comparison between early-absorbable and late-absorbable suture materials. World J Surg. 2000 Jun;24(6):747-51; discussion 752. doi: 10.1007/s002689910120. PMID 10773130
- [Background] Hodgson NC, Malthaner RA, Ostbye T. The search for an ideal method of abdominal fascial closure: a meta-analysis. Ann Surg. 2000 Mar;231(3):436-42. doi: 10.1097/00000658-200003000-00018. PMID 10714638
- [Background] Weiland DE, Bay RC, Del Sordi S. Choosing the best abdominal closure by meta-analysis. Am J Surg. 1998 Dec;176(6):666-70. doi: 10.1016/s0002-9610(98)00277-3. PMID 9926810
- [Background] Schumpelick V, Kingsanorth AN. Incisional Hernia. Questionnaire Survetta Meeting, March 1998: 496
- [Background] Schumpelick V, Arlt G, Klinge U. Versorgung von Nabelhernien und Narbenhernien. Dt. Aerzteblatt 94, 51-52. Dez. 1997 (35)
- [Background] Knaebel HP, Koch M, Sauerland S, Diener MK, Buchler MW, Seiler CM; INSECT Study Group of the Study Centre of the German Surgical Society. Interrupted or continuous slowly absorbable sutures - design of a multi-centre randomised trial to evaluate abdominal closure techniques INSECT-trial [ISRCTN24023541]. BMC Surg. 2005 Mar 8;5:3. doi: 10.1186/1471-2482-5-3. PMID 15755324
- [Background] Fischer L, Baumann P, Husing J, Seidlmayer C, Albertsmeier M, Franck A, Luntz S, Seiler CM, Knaebel HP. A historically controlled, single-arm, multi-centre, prospective trial to evaluate the safety and efficacy of MonoMax suture material for abdominal wall closure after primary midline laparotomy. ISSAAC-Trial [NCT005725079]. BMC Surg. 2008 Jul 21;8:12. doi: 10.1186/1471-2482-8-12. PMID 18644124
- [Background] Odermatt EK, Funk L, Bargon R, Martin DP, Rizk S, Williams SF. MonoMax Suture: A New Long-Term Absorbable Monofilament Suture Made from Poly-4-Hydroxybutyrate. International Journal of Polymer Science Volume 2012, Article ID 216137, 12 pages. doi:10.1155/2012/216137
- [Result] Albertsmeier M, Seiler CM, Fischer L, Baumann P, Husing J, Seidlmayer C, Franck A, Jauch KW, Knaebel HP, Buchler MW. Evaluation of the safety and efficacy of MonoMax(R) suture material for abdominal wall closure after primary midline laparotomy-a controlled prospective multicentre trial: ISSAAC [NCT005725079]. Langenbecks Arch Surg. 2012 Mar;397(3):363-71. doi: 10.1007/s00423-011-0884-6. Epub 2011 Dec 20. PMID 22183105
- [Result] Fink C, Baumann P, Wente MN, Knebel P, Bruckner T, Ulrich A, Werner J, Buchler MW, Diener MK. Incisional hernia rate 3 years after midline laparotomy. Br J Surg. 2014 Jan;101(2):51-4. doi: 10.1002/bjs.9364. Epub 2013 Nov 26. PMID 24281948